CLINICAL TRIAL: NCT05933382
Title: Investigation of the Effects of Mobilization With Movement Technique and Corticosteroid Injection on Pain, Functionality, and Proprioception in Rotator Cuff Lesions
Brief Title: Investigation of the Effects of Mulligan Mobilization and Corticosteroid Injection in Rotator Cuff Lesions
Acronym: Mobilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, burak menek, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MedipolPTR
Record Dates: First submitted 2023-06-12; First posted 2023-07-06 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Rotator Cuff Tears
Keywords: Mobilization with movement; Rotator cuff; Corticosteroid
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corticosteroid Group (Experimental): A conventional treatment program will be applied to individuals in both groups 5 days a week for 3 weeks. The conventional exercise program will consist of wand exercises, Codman exercises, stretching exercises for all ranges of motion, and TENS (100Hz, 15 minutes). A corticosteroid injection will be administered to the shoulder region of the first group prior to treatment.
  Interventions: Other: Corticosteroid Group
- Mulligan Group (Experimental): A conventional treatment program will be applied to individuals in both groups 5 days a week for 3 weeks. The conventional exercise program will consist of wand exercises, Codman exercises, stretching exercises for all ranges of motion, and TENS (100Hz, 15 minutes). In addition to the conventional treatment program, a mobilization technique with movement will be applied twice a week, with 10 repetitions.
  Interventions: Other: Mulligan Group

INTERVENTIONS:
Other: Corticosteroid Group — Conventional exercise and corticosteroid injection
  Arms: Corticosteroid Group
Other: Mulligan Group — Conventional exercise and mulligan mobilization
  Arms: Mulligan Group

SUMMARY:
Chronic shoulder pain, predominantly caused by rotator cuff disorders represents one of the most frequently encountered musculoskeletal issues within the community. Rotator cuff tears are a crucial pathophysiological contributor to shoulder pain. Individuals afflicted with this condition frequently report nocturnal intensification of pain and movement-specific aggravation, especially during overhead activities. The condition is frequently correlated with functional impairment, with many patients noting a sensation of weakness. Conservative treatment of the rotator cuff tear consists of a wide range of procedures such as exercise therapy; and/or local anesthetic, ice/heat therapy, electrotherapy, various types of manual therapy and joint mobilization procedures. Corticosteroid injection approach is an alternative method to these applications The subacromial corticosteroid injection is an intervention technique that has been utilized for short-term relief over numerous years.Given the restricted self-repair capabilities of tendons the consideration of novel biological treatment strategies for tendinopathies has gained prominence in recent times. Nonetheless, there remains a lack of sufficient scientific evidence to substantiate their efficacy.Mulligan mobilization techniques are manual therapy techniques that aim to increase normal joint movement and reduce pain levels by correcting the biomechanical structure of joint surfaces to provide a pain-free range of motion. A review of the literature reveals no studies comparing the Mulligan mobilization technique and corticosteroid injections in rotator cuff tears. The aim of our study is to examine the effects of the Mulligan mobilization technique and corticosteroid injections on pain, range of motion, functionality and proprioception in individuals with rotator cuff tears.

DETAILED DESCRIPTION:
Individuals diagnosed with rotator cuff rupture presenting at Medipol Esenler Hospital will be included in the study. Participants will be randomly divided into 2 groups. A conventional treatment program will be applied to individuals in both groups 5 days a week for 3 weeks. The conventional exercise program will consist of wand exercises, Codman exercises, stretching exercises for all ranges of motion, and TENS (100Hz, 15 minutes). A corticosteroid injection will be administered to the shoulder region of the first group prior to treatment. For the second group, in addition to the conventional treatment program, a mobilization technique with movement will be applied twice a week, with 10 repetitions. Inclusion Criteria:

* Being between the ages of 40 and 60
* Not having had any shoulder surgery before
* Having been diagnosed with a rotator cuff lesion
* Not having any orthopedic or cardiac problems that could hinder participation in the study and evaluation

Exclusion Criteria:

* Having a pathology affecting the shoulder area
* Having had any shoulder surgery
* Individuals who are non-cooperative or have mental problems
* Individuals with neurological, cardiac, and vascular problems
* Individuals who have participated in any physiotherapy program directed towards the shoulder in the last three months

Evaluation Scales to be Used:

* Visual Analog Scale - VAS
* Joint Range of Motion - Becure extremity ROM
* Joint Position Sense - Becure extremity ROM
* Disability of the Arm, Shoulder and Hand Questionnaire - DASH

Evaluation Methods:

1. Visual Analog Scale (VAS) The Visual Analog Scale is a commonly preferred evaluation method in the clinic and literature studies for measuring pain intensity. Patients' pain levels are determined by numbering 0-10. 0 indicates no pain, and 10 represents the most severe pain experienced.
2. Joint Range of Motion The normal joint range of motion was evaluated with the Becure Extremity ROM. Becure Extremity ROM is a system that allows for the objective measurement of joint range of motion by using its camera and sensors to detect reference points during extremity movements. In the Becure Extremity ROM system, the patient is expected to stand in front of the camera and perform the movement to be measured. In our study, the shoulder joint's flexion, extension, abduction, internal and external rotation ranges of motion were evaluated in degrees with Becure Extremity ROM.
3. Joint Position Sense The joint position sense measurements of the individuals participating in the study will be evaluated with a goniometer. Individuals will be asked to lift their shoulder to a certain degree, and then bring it back to the same angle value with their eyes closed. The angle value formed when eyes are open and closed will be recorded, and the difference between shoulder angles will be calculated. Joint position sense will be applied at 30 and 60 degrees of flexion and abduction movements.
4. Disability of the Arm, Shoulder, and Hand Questionnaire (DASH) The DASH, developed as a result of the collaboration of the American Academy of Orthopedic Surgeons and other groups, is a scale that evaluates physical restrictions and function in upper extremity lesions[18]. The DASH questionnaire consists of three subsections. The first part contains 30 questions; 21 questions evaluate the difficulties encountered in the patient's daily life functions, 5 questions are about symptoms, and the other 4 questions assess social life, work, sleep, and the individual's self-confidence. The part with 4 questions (optional Work Module (DASH- FS)) measures the difficulties encountered in the individual's work life.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Being between the ages of 40 and 60
* Not having had any shoulder surgery before
* Having been diagnosed with a rotator cuff lesion
* Not having any orthopedic or cardiac problems that could hinder participation in the study and evaluation

Exclusion Criteria:

Exclusion Criteria:

* Having a pathology affecting the shoulder area
* Having had any shoulder surgery
* Individuals who are non-cooperative or have mental problems
* Individuals with neurological, cardiac, and vascular problems
* Individuals who have participated in any physiotherapy program directed towards the shoulder in the last three months

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Visuel Analogue Scale (VAS) | 5 minutes
  The score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Normal range of motion and proprioception | 10 minutes
  Normal range of motion and proprioception can be measured with Becure Extremity ROM

SECONDARY OUTCOMES:
Functionality | 5 minutes
  Arm, Shoulder and Hand Problems Survey

CONTACTS AND LOCATIONS:
Overall Officials: Merve YILMAZ MENEK, PhD, Study Director — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Menek B, Menek MY. The efficacy of Mulligan mobilization and corticosteroid injection on pain, functionality, and proprioception in rotator cuff tears: A randomized controlled trial. J Hand Ther. 2025 Jul-Sep;38(3):410-417. doi: 10.1016/j.jht.2024.12.016. Epub 2025 Feb 6. PMID 39919923